CLINICAL TRIAL: NCT00410826
Title: Multicenter Randomized Phase II Study of Erlotinib, Cisplatin and Radiotherapy Versus Cisplatin and Radiotherapy in Patients With Stage III and IV Squamous Cell Carcinoma of the Head and Neck
Brief Title: Cisplatin and Radiation Therapy With or Without Erlotinib Hydrochloride in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Renato Martins, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6106; NCI-2009-01546 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT01009489 (obsolete NCT alias)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride; Cisplatin; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (chemo, radiotherapy, enzyme inhibitor/radiosensitizer) (Experimental): Patients receive cisplatin IV on days 1, 22, and 43 and undergo 3-dimensional conformal or intensity modulated radiotherapy once daily, 5 days per week, on days 1-47. Patients also receive erlotinib hydrochloride PO once daily on days -7 to 47.
  Interventions: Drug: erlotinib hydrochloride; Drug: cisplatin; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy; Procedure: quality-of-life assessment
- Arm II (chemotherapy, radiotherapy) (Active Comparator): Patients receive cisplatin and radiotherapy as in Arm I.
  Interventions: Drug: cisplatin; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
  Arms: Arm I (chemo, radiotherapy, enzyme inhibitor/radiosensitizer)
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Radiation: 3-dimensional conformal radiation therapy — 35 fractions
  Other Names: 3D-CRT; conformal radiation therapy
Radiation: intensity-modulated radiation therapy — 35 fractions
  Other Names: IMRT
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized phase II trial is studying cisplatin and radiation therapy together with or without erlotinib hydrochloride to compare how well they work in treating patients with stage III or stage IV head and neck cancer. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also make tumor cells more sensitive to radiation therapy. Giving cisplatin and radiation therapy together with erlotinib hydrochloride may kill more tumor cells. It is not yet known whether cisplatin and radiation therapy are more effective with or without erlotinib hydrochloride in treating head and neck cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the complete response rate in patients with locally advanced head and neck cancer, treated with cisplatin, radiotherapy and erlotinib (erlotinib hydrochloride) versus cisplatin and radiotherapy alone.

SECONDARY OBJECTIVES:

I. Evaluate whether the addition of erlotinib increases the acute and long term toxicities of cisplatin and radiotherapy, in patients with locally advanced head and neck cancer.

II. Compare the disease-free and overall survivals of patients with locally advanced head and neck cancer treated with cisplatin and radiotherapy, with and without erlotinib.

III. Evaluate whether the symptomatic improvement observed in the first week of erlotinib alone predicts for complete response and long term disease control.

IV. Correlate epidermal growth factor receptor (EGFR), p16 and excision repair cross-complementing 1 (ERCC-1) expression with response outcome to therapy with cisplatin and radiation with and without erlotinib.

V. Identify other molecular correlates that may be relevant in the pathogenesis of squamous cell carcinoma of head and neck (SCCHN) or response to therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cisplatin intravenously (IV) on days 1, 22, and 43 and undergo 3-dimensional conformal or intensity modulated radiotherapy once daily, 5 days per week, on days 1-47. Patients also receive erlotinib hydrochloride orally (PO) once daily (QD) on days -7 to 47.

ARM II: Patients receive cisplatin and undergo radiotherapy as in Arm I.

Within 10-14 weeks after completion of study treatment, patients with N2 or N3 disease at the time of screening undergo a neck dissection.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or pathological documented squamous cell carcinoma of oral cavity, oropharynx, larynx, and hypopharynx; patients with nasopharyngeal carcinoma can be included if the patients have grades I or II tumors according to the World Health Organization (WHO) classification
* Stage III or IV according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual, Sixth Edition (2002)
* Unresectable or resection with significant morbidity
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measurable Disease, defined according to Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
* Bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x ULN
* Calculated creatinine clearance >= 55ml/min (using the Cockcroft-Gault formula)
* Platelet count >= 100 x 10^9 /L
* Absolute neutrophil count (ANC) >= 1.25 x 10^9 /L
* Signed informed consent
* Male and female patients with reproductive potential must use an acceptable contraceptive method
* Authorization from a dentist to begin radiation therapy

Exclusion Criteria:

* Second primary malignancy that is clinically detectable or clinically significant at the time of consideration for study enrollment
* Inability or unwillingness to comply with radiotherapy
* Evidence of clinically significant congestive heart failure; patients must be able to tolerate hydration required during cisplatin chemotherapy
* Diarrhea > grade 1 at the time of enrollment
* Prior radiotherapy, chemotherapy, or investigational treatment for squamous cell carcinoma of head and neck
* Prior treatment with an investigational or marketed inhibitor of the EGFR pathway
* Use of cytochrome P450 3A4 (CYP3A4) inducers
* Presence of systemic metastases (M1)
* Pregnant or breast-feeding women
* Known human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2006-06; Primary Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato Martins, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (9):
- United States (9):
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - University of New Mexico Health Science CCOP, Albuquerque, New Mexico
  - University of North Carolina, Chapel Hill, North Carolina
  - New Hanover Radiation Oncology Center, Wilmington, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Cancer Institute-Boston Cancer Group PLC, Memphis, Tennessee
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Multicare Health System, Tacoma, Washington

REFERENCES:
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165
- [Derived] Bauman JE, Austin MC, Schmidt R, Kurland BF, Vaezi A, Hayes DN, Mendez E, Parvathaneni U, Chai X, Sampath S, Martins RG. ERCC1 is a prognostic biomarker in locally advanced head and neck cancer: results from a randomised, phase II trial. Br J Cancer. 2013 Oct 15;109(8):2096-105. doi: 10.1038/bjc.2013.576. Epub 2013 Sep 24. PMID 24064970
- [Derived] Martins RG, Parvathaneni U, Bauman JE, Sharma AK, Raez LE, Papagikos MA, Yunus F, Kurland BF, Eaton KD, Liao JJ, Mendez E, Futran N, Wang DX, Chai X, Wallace SG, Austin M, Schmidt R, Hayes DN. Cisplatin and radiotherapy with or without erlotinib in locally advanced squamous cell carcinoma of the head and neck: a randomized phase II trial. J Clin Oncol. 2013 Apr 10;31(11):1415-21. doi: 10.1200/JCO.2012.46.3299. Epub 2013 Mar 4. PMID 23460709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized between December 2006 and October 2011.
Groups:
- Arm A (Cisplatin and Radiotherapy): Patients receive cisplatin IV on days 1, 22, and 43 and undergo 3-dimensional conformal or intensity modulated radiotherapy once daily, 5 days per week, on days 1-47.
- Arm B (Cisplatin, Radiotherapy, Erlotinib): Patients receive cisplatin and radiotherapy as in Arm A. Patients also receive erlotinib hydrochloride PO QD on days -7 to 47.
Period: Overall Study
Arm/Group | Arm A (Cisplatin and Radiotherapy) | Arm B (Cisplatin, Radiotherapy, Erlotinib)
Started | 105 | 99
Completed | 96 | 95
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Population: 204 patients were randomized. However, after completing study therapy, it became apparent that one participant had metastatic disease and was therefore, ineligible for study. This participant was excluded from subsequent results presented here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Cisplatin and Radiotherapy) | Arm B (Cisplatin, Radiotherapy, Erlotinib) | Total
Number analyzed (Participants) | 104 | 99 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 86 | 177
  >=65 years | 13 | 13 | 26
Age Continuous [Mean (Full Range); unit: years] | 57 [37 to 74] | 56 [35 to 77] | 56 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 8 | 28
  Male | 84 | 91 | 175
Region of Enrollment [Number; unit: participants]
  United States | 104 | 99 | 203

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Percentage of Participants With a Complete Response in Each Treatment Arm
Description: Complete response requires both a pathological complete response (independent of observer) and a complete response radiologically (RECIST 1.0).
Time Frame: 12 weeks after the completion of therapy
Measure: Number; unit: percentage of participants
Groups:
- Arm B (Cisplatin, Radiotherapy, Erlotinib): Patients receive cisplatin and radiotherapy as in Arm A. Patients also receive erlotinib hydrochloride PO daily on days -7 to 47.
Arm/Group | Arm A (Cisplatin and Radiotherapy) | Arm B (Cisplatin, Radiotherapy, Erlotinib)
Number analyzed (Participants) | 96 | 95
percentage of participants | 42 | 51

2. Secondary Outcome: Safety as Assessed Through Summaries of Adverse Events and Laboratory Test Results by Treatment Arm
Time Frame: 30 days after the completion of therapy
Reporting Status: Not Posted

3. Secondary Outcome: Progression Free Survival of Patients With Locally Advanced Head and Neck Cancer Treated With Cisplatin and Radiotherapy, With and Without Erlotinib Hydrochloride
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Every 3 months for up to 5 years
Measure: Number; unit: participants
Arm/Group | Arm A (Cisplatin and Radiotherapy) | Arm B (Cisplatin, Radiotherapy, Erlotinib)
Number analyzed (Participants) | 104 | 99
participants | 25 | 29

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the first day of study therapy through 30 days following the last day of study therapy.
Description: All grades of rash and pain were recorded. For all other adverse events, only grade 3 and higher events and events that led to a dose reduction or delay were recorded.
Arm/Group | Arm A (Cisplatin and Radiotherapy) | Arm B (Cisplatin, Radiotherapy, Erlotinib)
Serious Adverse Events (participants affected / at risk) | 32/96 | 38/95
Other Adverse Events (participants affected / at risk) | 87/96 | 91/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cisplatin and Radiotherapy) (N=96) | Arm B (Cisplatin, Radiotherapy, Erlotinib) (N=95)
hearing loss (Ear and labyrinth disorders) | 2 | 0
Cytopenias (Blood and lymphatic system disorders) | 2 | 1
nausea,vomiting, dehydration (Gastrointestinal disorders) | 7 | 16
mucositis, esophagitis (Gastrointestinal disorders) | 1 | 2
peritonitis, perforation (Gastrointestinal disorders) | 2 | 1
hyponatremia (Metabolism and nutrition disorders) | 2 | 1
elevated creatinine (Metabolism and nutrition disorders) | 3 | 5
pneumonia (Infections and infestations) | 2 | 3
Pulmonary embolism, deep vein thrombosis (Vascular disorders) | 3 | 2
mood alteration (Psychiatric disorders) | 1 | 1
Substance abuse, seizure (Psychiatric disorders) | 1 | 2
congestive heart disease, cardiac arrest (Cardiac disorders) | 1 | 3
Respiratory arrest, hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
renal failure (Renal and urinary disorders) | 2 | 0
tachycardia (Cardiac disorders) | 1 | 0
pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Cisplatin and Radiotherapy) (N=96) | Arm B (Cisplatin, Radiotherapy, Erlotinib) (N=95)
dermatitis, rash (Skin and subcutaneous tissue disorders) | 10 | 65
pain (Gastrointestinal disorders) | 54 | 50
mucositis, nausea, vomiting, dehydration (Gastrointestinal disorders) | 31 | 28
Cytopenias (Blood and lymphatic system disorders) | 23 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No